CLINICAL TRIAL: NCT05425602
Title: A I / II Clinical Study to Evaluate the Safety, Tolerance, Pharmacokinetic Characteristics and Efficacy of MAX-40279 (Multi-target Tyrosine Kinase Inhibitor) Combined With KN046 (Anti-PD-L1 / CTLA-4 Bispecific Antibody) in Patients With Advanced / Metastatic Solid Tumors
Brief Title: A Study of MAX-40279combined With KN046 in Patients With Advanced / Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAX-40279-007
Record Dates: First submitted 2022-04-18; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Advanced / Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAX40279-01+KN046 (Experimental): This is an open-label Phase I/II clinical study.
  Drug: Stage1: Dose1:MAX40279-01 (35mg BID)+KN046 ( 5mg/kg Q3Week)
  Drug: Stage1: Dose2:MAX40279-01( 50mg BID)+KN046 ( 5mg/kg Q3Week)
  Drug: Stage1: Dose3:MAX40279-01( 70mg BID)+KN046 ( 5mg/kg Q3Week)
  Drug: Stage2: Dose3:MAX40279-01( RP2D BID)+KN046 ( 5mg/kg Q3Week)
  Interventions: Drug: MAX-40279-01: 50mg/70mg

INTERVENTIONS:
Drug: MAX-40279-01: 50mg/70mg — [Stage 1]The starting dose of MAX-40279 was 35 mg BID, and three dose levels were initially set: 35 mg, 50 mg, and 70 mg administered twice daily (BID) continuously, and the dose of KN046 was 5 mg/kg as a fixed dose administered every 3 weeks. [Stage 2]When the RP2D dose is obtained in the dose-finding phase, the trial will enter the dose expansion phase.
  Other Names: KN046: 40mg/300mg

SUMMARY:
This include two parts, Stage 1 is a dose climbing study and Stage 2 is a dose extending study.

DETAILED DESCRIPTION:
This study is a study of MAX-40279 in patients with advanced / metastatic solid tumors. This study include two Parts, the Part 1 will assess the safety and efficacy of the dose climbing level of MAX-40279, and recommend a dose extending level of MAX-40279 for stage 2.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Males and/or females over age 18 and 75.
3. Histologically or cytologically documented local advanced / metastatic solid tumors who have failed standard treatment or cannot obtain standard treatment in the dose escalation stage; dose expansion stage group A: relapsed and refractory advanced gastric cancer; dose expansion stage group B: relapsed and refractory extensive stage small cell lung cancer; dose expansion stage group C: other relapsed and refractory solid tumors except group A
4. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Expected survival of more than 3 months.

Exclusion Criteria:

1. The adverse reactions of previous anti-tumor treatment have not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except alopecia and other adverse reactions without safety risks judged by the investigator)
2. Subject is known to have previous serious allergic reactions to macromolecular protein preparations/monoclonal antibodies, or known to any component of the test drug
3. Active systemic infectious diseases requiring intravenous antibiotic treatment 2 months before the first medication
4. Subject has poorly controlled cardiovascular and cerebrovascular clinical symptoms or diseases, including but not limited to: such as: (1) NYHA class II or higher heart failure or LVEF < 50%; (2) unstable angina pectoris; (3) myocardial infarction and cerebral infarction within 6 months; (4) clinically significant supraventricular or ventricular arrhythmias are still poorly controlled without clinical intervention or clinical intervention
5. brain metastases, spinal cord compression, carcinomatous meningitis with clinical symptoms, or other evidence of uncontrolled brain and spinal cord metastases, Patients who are not suitable by the investigator's judgment
6. Patients who have experienced ≥ grade 3 immune-related adverse events in immunotherapy (except grade 3 hypothyroidism that can be controlled by drugs)
7. Patients who have other malignant tumors within 5 years before enrollment,Exceptions: a. radical cervical carcinoma in situ or non-melanoma skin cancer; b. radical second primary cancer without recurrence within five years; c. the investigator believes that the double primary cancer can benefit from this study; d. the investigator has clearly excluded which primary tumor source the metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
DLT | through study Stage1 completion，an average of 6 months
Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) | through study Stage1 completion，an average of 6 months
ORR | through study Stage2 completion，an average of 24 months
PFS | through study Stage2 completion，an average of 24 months
Adverse events (AEs), serious adverse events (SAEs) | through study Stage2 completion，an average of 24 months
laboratory tests | through study Stage2 completion，an average of 24 months
vital signs | through study Stage2 completion，an average of 24 months
12 ECG | through study Stage2 completion，an average of 24 months
physical examination abnormalities | through study Stage2 completion，an average of 24 months

SECONDARY OUTCOMES:
Adverse events (AEs), serious adverse events (SAEs) | through study Stage1 completion，an average of 6 months
Cmax | through study Stage1 completion，an average of 6 months
Anti-KN046 antibody (ADA | through study Stage1 completion，an average of 6 months
Duration of response (DOR) Overall survival (OS); Anti-KN046 antibody (ADA); Plasma concentrations of MAX-40279 and KN046 [Stage 2] | through study Stage2 completion，an average of 24 months
(AUC0-t and AUC0-t, ss) | through study Stage1 completion，an average of 6 months
Tmax | through study Stage1 completion，an average of 6 months
Overall response rate (ORR) | through study Stage1 completion，an average of 6 months
disease control rate (DCR) | through study Stage1 completion，an average of 6 months
duration of response (DOR) | through study Stage1 completion，an average of 6 months
progression-free survival (PFS) | through study Stage1 completion，an average of 6 months
overall survival (OS) | through study Stage1 completion，an average of 6 months
DcR | through study Stage2 completion，an average of 24 months
DoR | through study Stage2 completion，an average of 24 months
OS | through study Stage2 completion，an average of 24 months
Anti-KN046 antibody (ADA) | through study Stage2 completion，an average of 24 months
Rac (AUC0-t, ss/AUC0-t) | through study Stage1 completion，an average of 6 months
laboratory tests | through study Stage1 completion，an average of 6 months
vital signs | through study Stage1 completion，an average of 6 months
12 ECG | through study Stage1 completion，an average of 6 months
physical examination abnormalities | through study Stage1 completion，an average of 6 months

OTHER OUTCOMES:
FGFR1OP2-related protein expression levels and mutations, PD-L1 and related inflammatory factors correlate with efficacy [Stage 1] | through study Stage1 completion，an average of 6 months
FGFR1OP2-related protein expression levels and correlation of mutations, PD-L1, tumor mutation burden, and related inflammatory factors with efficacy.[ Stage 2] | through study Stage2 completion，an average of 24 months

IPD SHARING:
Plan to Share IPD: No